CLINICAL TRIAL: NCT05568251
Title: Transcranial Direct Current Stimulation Combined With Cognitive Training In Opioid Use Disorder
Brief Title: TDCS Combined With CT In Opioid Use Disorder
Acronym: OpiStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Research, Treatment and Training Center for Alcohol and Substance Dependence (AMATEM) (Unknown)
Responsible Party: Principal Investigator, Serkan Aksu, Assistant Proffessor Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-438
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Opioid Use Disorder
Keywords: brain stimulation; cognitive functions; neuropsychological evaluation; opioid use disorder; transcranial direct current stimulation
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS combined with Cognitive Training (Active Comparator)
  Interventions: Device: transcranial Direct Current Stimulation; Procedure: Cognitive training
- Sham tDCS combined with Cognitive Training (Sham Comparator)
  Interventions: Device: transcranial Direct Current Stimulation; Procedure: Cognitive training

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — Participants will receive a single session of active/sham tDCS. During each session, 2 milliAmpers of active or sham tDCS will be applied for 20 minutes over the dorsolateral prefrontal cortex (right anodal/left cathodal).
Procedure: Cognitive training — Participants will be administered Game of Dice Task concurrent with the tDCS session

SUMMARY:
The aim of the present study is to investigate the effect of prefrontal transcranial Direct Current Stimulation (tDCS) combined with cognitive training on cognitive functions in individuals with Opioid Use Disorder (OUD). The participants will be allocated into active/sham groups (1:1) and will receive a single session of prefrontal tDCS combined with cognitive training. Outcomes of the active and sham groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 18-65 years
* being in the maintenance phase of the OUD treatment
* naivety to tDCS
* at least 5 years of education

Exclusion Criteria:

* current diagnosis of major depressive disorder
* current diagnosis or history of bipolar disorders, psychotic disorders, neurocognitive disorders, pervasive developmental disorders, mental retardation, severe neurological disorders,
* common tDCS contraindications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in the Iowa Gambling Task net score | Before and immediately after the intervention
  Iowa Gambling Task net score is the total score of the task (between -100 and 100) that generally assesses the decision making under ambiguity, but also assesses the decision making under risk at the later stages. Higher scores in the task represents better decision making and healthy people generally have scores above 8-10 in the task.
Changes in the Adjusted Number of Pumps in the Balloon Analogue Risk Task | Before and immediately after the intervention
  The Balloon Analogue Risk Task is the commonly used computerized measure of decision making under risk. Main outcome variable of the task is the Adjusted Number of Pumps which includes the mean number of pumps in the trials that not resulted with an explosion. Lower values mean lower impulsivity.

SECONDARY OUTCOMES:
Changes in Interference Time in the Stroop Test | Before and immediately after the intervention
  The stroop effect (Interference Time) consists of both the semantic and the response conflict. Response conflict (time in milliseconds) is obtained by subtracting the semantic conflict (time in milliseconds obtained in the second step of the protocol) from the stroop effect (time in milliseconds obtained in the first step of the protocol). Minimum time difference is 0 and maximum time difference is 100 milliseconds. Lower time differences indicate better performance and higher time differences indicate worse performance.
Changes in the Stop Signal Reaction time in the Stop Signal Test | Before and immediately after the intervention
  The Stop-Signal Task (SST) is a task requiring inhibition of a prepotent motor response. The SST requires participants to respond to a target stimulus as quickly and accurately as possible by pressing a button, but also to withhold their response when they hear an auditory signal. Thus, this task involves a competition between activating and inhibiting processes. The primary outcome variable is change in the stop signal reaction time (SSRT) for the task administered seconds to minutes before and seconds to minutes after stimulation. The theoretical minimum is zero seconds and there is no theoretical maximum. Higher SSRT scores reflect greater impulsivity.
Changes in the verbal fluency performance | Before and immediately after the intervention
  Verbal fluency is a test that measure multiple domains of cognition such as executive functions and language functions. Phonemic Fluency assesses the number of words beginning with certain letters that participants can generate within 60 seconds, the semantic Fluency assesses the number of words within particular categories participants can generate within 60 seconds. Alternating fluency assesses the number of fruit-name pairs reported in a minute duration. Theoretical minimum is zero and there is no theoretical maximum . Lower scores indicate worse performance and higher scores indicate better performance.
Changes in the digit span performance | Before and immediately after the intervention
  The Digit Span test is a measure of verbal short-term/working memory. Subjects must recall all digits either in forward (digit span forward) or backward (digit span backward) order.
  Digit span forward total score: 0-10; higher score indicate better performance, digit span backwards total score: 0-10; higher score indicate better performance
Changes in the Trail Making Test A Time | Before and immediately after the intervention
  Trail Making A Test is a widely used as a quick and easy to administer measure of attention. Lower reaction times indicate better performance and higher reaction times indicate worse performance. Minimum time is 10 milliseconds and maximum time is 150 milliseconds.
Changes in the Trail Making Test B Time | Before and immediately after the intervention
  Trail Making B Test is a widely used as a quick and easy to administer measure of executive functions. Lower reaction times indicate better performance and higher reaction times indicate worse performance. Minimum time is 10 milliseconds and maximum time is 150 milliseconds.
Changes in the Letter Number Sequencing (LNS) Test performance | Before and immediately after the intervention
  Letter number is a test of working memory which involves ordering a series of up to 8 letters and numbers in which the numbers are repeated back first in order starting with the lowest number, then followed by the letters in alphabetical order. LNS consists of 10 items and each item has 3 trials rated as Incorrect (0) or Correct (1). The LNS total raw score (range 0 to 30) is auto-calculated by summing the 10 individual item scores (range 0 to 3 for each item). Higher number of correct items correlated to better performance and a negative change from baseline indicates worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Aksu, Principal Investigator — Istanbul University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul
  - Research, Treatment and Training Center for Alcohol and Substance Dependence (AMATEM), Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aksu S, Soyata AZ, Seker S, Akkaya G, Yilmaz Y, Kafali T, Evren C, Umut G. Transcranial direct current stimulation combined with cognitive training improves decision making and executive functions in opioid use disorder: a triple-blind sham-controlled pilot study. J Addict Dis. 2024 Apr-Jun;42(2):154-165. doi: 10.1080/10550887.2023.2168991. Epub 2023 Mar 2. PMID 36861945